CLINICAL TRIAL: NCT00285935
Title: Neurosteroid Metabolism and the Antidepressant Effects of Serotonin Specific Reuptake Inhibitors (SSRI's)
Brief Title: Cellular Aging and Neurobiology of Depression Study
Acronym: CAN-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-00825; R01MH083784 (NIH); K08MH126192 (NIH)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Neurobiology; Selective Serotonin Reuptake Inhibitor; SSRI; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with SSRI (Experimental): Depressed participants will receive 8 weeks of treatment with one of the following serotonin-specific reuptake inhibitors:
  fluoxetine (Prozac®), sertraline (Zoloft®), citalopram (Celexa®), escitalopram (Lexapro®)
  The specific drug used for treatment will be selected by the study clinician based on clinical interviews and the participants preferences. Participants will be monitored for response and side effects by study clinician and will return after 8 weeks for a follow up study visit.
  Interventions: Other: Standard Clinical Care with an SSRI

INTERVENTIONS:
Other: Standard Clinical Care with an SSRI — Participants who enroll in this phase are treated with an FDA-approved SSRI in an open-label "treatment-as-usual" manner, in accordance with clinical practices and at a titration rate no more rapid than the manufacturer's recommendations. The duration of the treatment phase is 8 weeks.
  Other Name: fluoxetine (Prozac®), Sertraline (Zoloft®), citalopram (Celexa®), escitalopram (Lexapro®)

SUMMARY:
We are conducting an eight week longitudinal study to learn if blood levels of certain naturally occurring compounds and genetic markers differ between patients with depression and healthy adults who are not depressed, and if any such differences relate to memory performance, mood, and neurobiology. We are also interested in how the gut microbiome is affected by antidepressant treatment.

We will do this by comparing the unmedicated depressed patients with matched healthy controls at baseline and then following the depressed patients over the course of eight weeks of standardized antidepressant treatment to gauge which baseline abnormalities normalize over the course of treatment.

DETAILED DESCRIPTION:
Following an initial telephone screen to assess inclusion and exclusion criteria, the evaluation will continue with an in-person screening evaluation to assess the presence or absence of active medical history and history of major psychiatric illness, as well as review of the consent document. If found to be eligible, participants would then be admitted to the study.

The next step for eligible, consenting depressed subjects and is a baseline visit. The baseline visit will last up to 3.5 hours. We will begin the baseline visit by collecting a urine sample for a drug (and, for women, pregnancy) test. As long as that is negative, we will then collect a blood sample of about 180 cc. After the blood draw, participants will complete cognitive tests and meet again with the study psychiatrist. Eligible consenting healthy controls will come in for a one time study visit and complete the same tests performed during the depressed subject baseline visit. Both depressed participants and healthy controls will return a stool sample collected at home with a kit given during the screening visit.

After the baseline visit, depressed subjects (but not healthy controls) will begin taking an FDA approved antidepressant, as prescribed by the study psychiatrist, for the next 8 weeks while they are enrolled in the study. The specific drug will be decided upon between the participant and the study psychiatrist at the in-person screening visit.

After 4 weeks, depressed participants will return to UCSF to meet again with the psychiatrist to discuss symptoms and how to continue treatment. They will be given an at home collection kit to return a stool sample at the last study visit.

4 weeks later (after 8 weeks in total), depressed participants will come back for an additional visit that will include the same blood draw and testing as the baseline visit. They also will return their stool sample. A physician-investigator will meet with the depressed subjects to review their clinical responses to treatment and to make further treatment suggestions, which the subjects may use in discussions of their future treatment options with their personal physicians. If a decision is made to discontinue antidepressant treatment, the subjects will be given instructions on how to withdraw from the medication, and will be given up to a 4 week supply of the drug to facilitate this withdrawal.

ELIGIBILITY:
All participants must meet the following criteria:

* Age 21-60 and able to give informed consent.
* Not "needle phobic," by self-report.
* English-speaking (to allow accurate use of behavioral rating scales and verbal cognitive tests).
* Females of child-bearing capacity must be non-pregnant (confirmed by urine pregnancy test) and using effective non-hormonal birth control (e.g. abstinence, condoms, IUD).
* Good general medical health; no significant uncontrolled illnesses that will invalidate the designated outcome measures.
* Clinical labs (electrolytes, liver function test, CBC) with no clinically significant abnormalities that result in medical treatment that will invalidate the designated outcome measures.
* Negative urine toxicology (drugs of abuse) screen.
* Taking no medication or drugs likely to interfere with the study objectives (including statins or medications that affect hormones [e.g. birth control pills or steroids]).
* Free of all psychotropic medications (including antidepressants) for at least 6 weeks (with the exception of prn short-acting benzodiazepines or sedative-hypnotics, < 3 doses per week, and none for 5 drug half-lives before the study).
* No vaccines for at least 4 weeks prior to baseline blood draw (including the flu shot).
* Not currently anemic (Hct of 36-48 for females and 38-54 for males, or Hgb of 12.5-20) and has not donated blood for at least 8 weeks prior to baseline blood draw.
* No neurological disorders and no history of concussion with a black-out that lasted > 10 minutes.
* Willing to provide stool sample

Additional criteria for Depressed Participants:

* Current DSM-5 diagnosis of Major Depressive Disorder, unipolar, with non-psychotic features.
* Baseline 17-item Hamilton Depression Rating Scale (HDRS) rating of >= 17, or Baseline 25-item HDRS rating of >= 20.
* Current depressive episode duration of > 6 weeks.
* No current, active suicidal intent; HDRS "suicidality" item rating <= 2 OR by clinician determination.
* No recent (< 6 month) history of substance or alcohol use disorder(s), with the exception of tobacco use (DSM-5 criteria).
* No current (in the last month) diagnosis of Post-Traumatic Stress Disorder (DSM-5 criteria).
* No anticipated changes in psychotherapeutic interventions during the course of the study.

Additional criteria for Normal Controls:

• No history of DSM-5 Axis I diagnoses

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2010-12-16 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Depression ratings at baseline and Week 8 | baseline and Week 8
Serum levels of steroids and neurosteroids at baseline and Week 8 | baseline and Week 8

SECONDARY OUTCOMES:
Serum levels of oxidative stress markers at baseline and Week 8 | baseline and Week 8
Serum levels of cytokines and immune markers at baseline and Week 8 | baseline and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Owen Wolkowitz, MD, Principal Investigator — University of California, San Francisco; Ryan Rampersaud, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rampersaud R, Wu GWY, Reus VI, Lin J, Blackburn EH, Epel ES, Hough CM, Mellon SH, Wolkowitz OM. Shorter telomere length predicts poor antidepressant response and poorer cardiometabolic indices in major depression. Sci Rep. 2023 Jun 23;13(1):10238. doi: 10.1038/s41598-023-35912-z. PMID 37353495
- [Derived] Rampersaud R, Protsenko E, Yang R, Reus V, Hammamieh R, Wu GWY, Epel E, Jett M, Gautam A, Mellon SH, Wolkowitz OM. Dimensions of childhood adversity differentially affect biological aging in major depression. Transl Psychiatry. 2022 Oct 4;12(1):431. doi: 10.1038/s41398-022-02198-0. PMID 36195591
- [Derived] Wolkowitz OM, Mellon SH, Epel ES, Lin J, Reus VI, Rosser R, Burke H, Compagnone M, Nelson JC, Dhabhar FS, Blackburn EH. Resting leukocyte telomerase activity is elevated in major depression and predicts treatment response. Mol Psychiatry. 2012 Feb;17(2):164-72. doi: 10.1038/mp.2010.133. Epub 2011 Jan 18. PMID 21242992